CLINICAL TRIAL: NCT02033473
Title: Effect of Apelin on Insulin Sensitivity: Proof of Concept in Healthy Volunteers
Acronym: APELINS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 13 182 03; HAO 2013 (Other: Hors Appel d'Offres)
Record Dates: First submitted 2013-12-12; First posted 2014-01-10 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Healthy
Keywords: Apelin; insulin; volunteers
MeSH Terms: conditions — Insulin Resistance | interventions — Apelin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apelin (Experimental): An apelin clamp in which an apelin infusion will be administered prior to reference clamp
  Interventions: Drug: Apelin; Drug: Placebo
- Placebo (Placebo Comparator): A clamp reference during which a placebo solution (saline solution) will be administered prior to apelin clamp
  Interventions: Drug: Apelin; Drug: Placebo

INTERVENTIONS:
Drug: Apelin — An apelin clamp in which an apelin infusion will be administered
Drug: Placebo — A clamp reference during which a placebo solution (saline solution) will be administered

SUMMARY:
The (PYR1)-apelin-13 is an endogenous peptide discovered relatively recently (1998). The apelin and its receptor, which is named apj, are expressed in many tissues including sensitive to the action of insulin, such as skeletal muscle, adipose tissue and heart tissue.

Recent work by the team of Prof. P.Valet (INSERM U1048, Toulouse) opened a new field of investigation, demonstrating for the first time in mouse models that apelin exerts a glucose-regulating in vivo action. The investigators propose a translational clinical research project whose goal is to provide the proof of concept of the favorable influence of apelin on insulin sensitivity in humans.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 to 40 years.
* BMI between 25 and 30 kg / cm ² (excluding terminals).
* Free of known chronic disease and any medication (any medication within 30 days prior to the inclusion visit).
* Non-pathological ECG.
* Heart rate between 50 and 80 beats per minute rest.
* Complete Blood Count (CBC) with no significant anomaly in terms of the investigator.
* Liver function tests without clinically significant abnormalities in terms of the investigator.
* Renal function tests without clinically significant abnormalities in terms of the investigator.
* Serum electrolytes without clinically significant abnormalities in terms of the investigator.
* Fasting plasma glucose less than 1.1 g / l.
* HbA1c within the normal range (4-6%).
* Good peripheral vein (forearm and back of the hand).
* Agreement to participate in the establishment of a serum bank.
* Sedentary or practicing occasional physical activity.
* Ability to sign informed consent.
* Affiliation to a social security scheme.

Exclusion Criteria:

* Risk factor, treatment or ECG as recommended by International Conference on Harmonization E14 (ICH E14) "Clinical Evaluation of QT / corrected QT interval (QTc Interval= Prolongation and Proarrhythmic Potential for Non-Antiarrhythmic Drugs"
* Repeated a QTc interval> 450 ms measurement
* Risk factor: myocardial infarction, hypokalemia, family history of long QT syndrome
* Personal history of cancer.
* Positive HIV serology.
* Hepatitis B serology positive.
* Positive hepatitis C serology.
* Cognitive impairment or mental illness (at the discretion of the investigator).
* Chronic excessive alcohol consumption (consumption> 30g/jour or 210g/week).
* Person under judicial protection, guardianship.
* Subject with a resting systolic blood pressure greater than 140 mm Hg and diastolic blood pressure greater than 90 mmHg
* Smoking> 10 cig / day and can not be interrupted for 24 hours.
* Subject exclusion period of another protocol.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Rate of glucose infusion | The last 30 minutes of a hyperinsulinemic euglycemic clamp
  Measuring the difference between the rate of glucose infusion measured in the last 30 minutes of a hyperinsulinemic euglycemic clamp in the presence of a continuous infusion (PYR1)-apelin-13 infusion rate of glucose measured in the same conditions in the presence of a continuous infusion of placebo.

SECONDARY OUTCOMES:
Calculation of the index of insulin sensitivity (Si) | During 240 minutes at visits 2 and 3
Changes in the measurement of systolic blood pressure during each clamp | During 240 minutes at visits 2 and 3
Changes in the measurement of diastolic blood pressure during each clamp | During 240 minutes at visits 2 and 3
Changes in heart rate measurement during each clamp | During 240 minutes at visits 2 and 3
Changes in ECG during each clamp | During 240 minutes at visits 2 and 3
Clinical signs of intolerance / allergy / toxicity at visit 2,3 and 4 | During 240 minutes at visits 2 and 3
Determination of plasma insulin at all sampling | During 240 minutes at visits 2 and 3
Determination of plasma glucagon at all sampling times | During 240 minutes at visits 2 and 3
Determination of plasma apelin at all sampling times | During 240 minutes at visits 2 and 3
Determination of plasma leptin at all sampling times | During 240 minutes at visits 2 and 3
Determination of plasma adiponectin at all sampling times | During 240 minutes at visits 2 and 3

CONTACTS AND LOCATIONS:
Overall Officials: Pierre GOURDY, Md, PhD, Principal Investigator — University Hospital of Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France

REFERENCES:
- [Result] Gourdy P, Cazals L, Thalamas C, Sommet A, Calvas F, Galitzky M, Vinel C, Dray C, Hanaire H, Castan-Laurell I, Valet P. Apelin administration improves insulin sensitivity in overweight men during hyperinsulinaemic-euglycaemic clamp. Diabetes Obes Metab. 2018 Jan;20(1):157-164. doi: 10.1111/dom.13055. Epub 2017 Aug 10. PMID 28681996